CLINICAL TRIAL: NCT04967456
Title: Efficacy of Laser Doppler Flowmetry, as a Diagnostic Tool in Assessing Revascularization of Traumatised Teeth
Brief Title: Efficacy of Laser Doppler Flowmetry as a Diagnostic Tool in Assessing Revascularization of Traumatised Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Plovdiv Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MedicalUniversity_Doppler
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Trauma; Diagnosis Dual
Keywords: Laser Doppler flowmetry; pulpal blood flow; pulp vitality; traumatised teeth; paediatric dentistry
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: a randomized, split-mouth, controlled, clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Measurement of pulpal blood flow of traumatised tooth (Active Comparator): In the split-mouth design, the traumatised maxillary incisor will be investigated using Laser Doppler flowmetry.
  Interventions: Diagnostic Test: Measurement of pulpal blood flow of traumatised tooth
- Measurement of pulpal blood flow of non-traumatised tooth (Other): In the split-mouth design, this arm - the non-traumatised maxillary incisor, contralateral tooth, will be investigated using Laser Doppler flowmetry as a control tooth.
  Interventions: Diagnostic Test: Measurement of pulpal blood flow of traumatised tooth

INTERVENTIONS:
Diagnostic Test: Measurement of pulpal blood flow of traumatised tooth — Measurement of the blood flow of the dental pulp will be performed, using a laser doppler flow monitor "mVMS-LDF2TM" (Moor Instruments Ltd Millwey Axminster Devon, UK), emission wavelength 785nm±10nm, dual-channel laser Doppler monitoring option. Two probes will be used, each consisting of one afferent and one efferent optic fiber to conduct the light to and from the tooth surface. The probe is stainless steel needle-like tube, which is 10-80 mm long and 1.5 mm in the diameter. The utilised parameter settings will be: Average power - 1.0 mV; Diameter of the probe - 1.5 mm; Frequency - 40 Hz; Monitoring time-180 seconds (sec)

SUMMARY:
The aim of the study is to evaluate the efficacy of Laser Doppler flowmetry in determining the changes in the pulpal blood flow during the post-traumatic period of traumatised permanent teeth.

DETAILED DESCRIPTION:
Traumatic injuries of permanent teeth in children and adolescents are very common. The conventional pulp vitality tests are inaccurate and unreliable techniques in assessing the pulp vitality during the post-traumatic period, as well as during the immature teeth examination. The aim is to evaluate the efficacy of Laser Doppler flowmetry in determining the changes in the pulpal blood flow during the post-traumatic period of traumatised permanent teeth. The study is designed as a randomized, split-mouth, controlled clinical trial. The measurement of the blood flow of the dental pulp of both, traumatised and non-traumatised teeth, will be performed, using a laser doppler flow monitor, emission wavelength 785nm±10nm, dual-channel laser Doppler monitoring option.

ELIGIBILITY:
Inclusion Criteria:

1. Fit and healthy subjects aged < 18-year-old;
2. Subjects with maxillary permanent incisor subjected to a traumatic injury without any dentoalveolar trauma involvement and have a contralateral homologous tooth with no signs/symptoms of injury;
3. Subjects attended their first dental visit within 3 days of the dental trauma;
4. Sensitivity value of the electric pulp test over 200 μA;
5. Subjects with at least one vital and non-traumatised maxillary incisor acting as a control tooth;
6. Ability to obtain a verbal acceptance from all the subjects to comply with all the treatments and follow-up timepoints attendance;
7. Ability to obtain written informed consent by the patients' parents/guardians for treatment, participation in the study and publication

Exclusion Criteria:

1. Subjects who were undergoing therapy for neurological conditions or with mental or cognitive problems;
2. Subjects who were taking sedative, analgesic, and/or anti-inflammatory medication 7 days prior to the treatment commencement;
3. Subjects who have never had any first dental visit or treatment;
4. Subjects with systemic diseases or physiological development delay;
5. Subjects with active infectious diseases such as; influenza, scarlet fever, etc.
6. Subjects with restorations covered more than half the labial surface of the investigated teeth.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-07-09 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Changes in pulpal blood flow | 180 seconds
  The traumatised and non-traumatised teeth, test and control, will be assessed by LDF, providing an accurate and precise investigation. The temperature in the dental office will be constant and the patient will be seated in a "state position" in the dental chair. According to the manufacturer's recommendations, a patient's relaxation of 10 minutes before the monitoring process will be obtained. The measurements of blood flow will be performed for 180 seconds at each session. All the measurements will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Shindova, PhD, Principal Investigator — Plovdiv Medical University
Locations (2):
- Bulgaria (2):
  - Department of Paediatric Dentistry, Faculty of Dental Medicine, Medical University - Plovdiv, Bulgaria, Plovdiv
  - Medical University - Plovdiv, Bulgaria, Plovdiv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Belcheva A, Shindova M, Hanna R. Efficacy of Laser Doppler Flowmetry, as a Diagnostic Tool in Assessing Pulp Vitality of Traumatised Teeth: A Split Mouth Clinical Study. J Pers Med. 2021 Aug 17;11(8):801. doi: 10.3390/jpm11080801. PMID 34442445